CLINICAL TRIAL: NCT07331480
Title: Combined Effect of Rhythmic Auditory Stimulation and Functional Electrical Stimulation on Gait in Children With Hemiparesiss
Brief Title: Combined Auditory and Functional Electrical Stimulation on Gait in Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Ibrahim, assistant professor of pediatric physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pediatrics physical therapy
Record Dates: First submitted 2025-12-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Hemiparesis
Keywords: auditory; electrical stimulation; gait
MeSH Terms: conditions — Paresis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: two groups control and study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): regular physical therapy exercises
  Interventions: Other: gait training; Other: Exercise; Other: control group gait training
- study group (Experimental): auditory and functional electrical stimulation effect on gait
  Interventions: Other: gait training; Other: Exercise; Other: control group gait training

INTERVENTIONS:
Other: gait training — use combination of auditory stimulation and functional electrical stimulation effect on gait training in children with hemiparesis
  Other Names: gait training for study group
Other: Exercise — gait training
Other: control group gait training — rehabilitation

SUMMARY:
Hemiparetic cerebral palsy has been characterized increased the asymmetry in the distribution of body weight between the affected and unaffected lower limbs and ineffective foot clearance during swing phase. This has been shown to result in an increased in the abnormal gait. This study aims to investigate the effect of rhythmic auditory stimulation combined with functional electrical stimulation on gait in children with hemiparetic cerebral palsy.

DETAILED DESCRIPTION:
A few studies have examined the benefits of music therapy showed that that weight-bearing stance time on the paretic side and stride symmetry improved with rhythmic cueing. Furthermore, the variability of integrated amplitude ratios decreased during the midstance/push off phase on the paretic side.

Improving walking safety, speed, postural control, balance and gait training are essential objectives for gait rehabilitation for hemiparetic children to prevent falls and subsequently to improve quality of life.

ELIGIBILITY:
Inclusion Criteria: hemiparesiss children aged 6 to 10 -

Exclusion Criteria: recent Botox or lower limb surgery

-

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
gait parameters | 3 months
  step length in cm

SECONDARY OUTCOMES:
range of motion | 3 months
  hip range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abbass, phd, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt